CLINICAL TRIAL: NCT01848990
Title: CONtinuous Subcutaneous Insulin Infusion STudy ENrolling Type 1 (CONSISTENT 1): Evaluation of Metabolic Outcomes and Safety of Hylenex Recombinant (Hyaluronidase Human Injection) Used as a Preadministration Infusion Site Treatment in Subjects With Type 1 Diabetes (T1DM) Using Continuous Subcutaneous Insulin Infusion (CSII)
Brief Title: CONSISTENT 1: Metabolic and Safety Outcomes of Hylenex Recombinant (Hyaluronidase Human Injection) Preadministered at CSII Infusion Site in Participants With Type 1 Diabetes Mellitus (T1DM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Halo-117-403
Record Dates: First submitted 2013-04-29; First posted 2013-05-08 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Sub Cutaneous Insulin Infusion; Rapid Acting Analog Insulin; Hylenex; Halozyme; Phase 4
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Akacid-medical-formulation; Insulin Lispro; Insulin Aspart; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Commercial Hylenex Recombinant (Formulation 1) (Experimental): Hylenex Formulation 1: For 6 months, participants received their regular treatment of rapid-acting continuous subcutaneous insulin infusion (CSII) (for example, insulin lispro, insulin aspart, and insulin glulisine). Additionally, during this 6-month treatment period, the participants received a pretreatment dose of the commercial form of Hylenex recombinant, delivered at 150 units (U) through their insulin infusion cannula each time they changed infusion sets (every 2 to 3 days).
  Interventions: Drug: Commercial Hylenex® recombinant (hyaluronidase human injection); Drug: Insulin lispro; Drug: Insulin aspart; Drug: Insulin glulisine
- Precommercial Hylenex Recombinant (Formulation 2) (Experimental): Hylenex Formulation 2: For 6 months, participants received their regular treatment of rapid-acting CSII (for example, insulin lispro, insulin aspart, and insulin glulisine). Additionally, during this 6-month treatment period, the participants received a pretreatment dose of the precommercial form of Hylenex recombinant, delivered at 150 units (U) through their insulin infusion cannula each time they changed infusion sets (every 2 to 3 days).
  Interventions: Drug: Precommercial Hylenex recombinant (hyaluronidase human injection); Drug: Insulin lispro; Drug: Insulin aspart; Drug: Insulin glulisine
- Standard Rapid-Acting Insulin CSII (Active Comparator): Participants received their regular treatment of rapid-acting CSII (for example, insulin lispro, insulin aspart, and insulin glulisine) for 6 months.
  Interventions: Drug: Insulin lispro; Drug: Insulin aspart; Drug: Insulin glulisine

INTERVENTIONS:
Drug: Commercial Hylenex® recombinant (hyaluronidase human injection)
  Other Names: Formulation 1; Hylenex; Recombinant human hyaluronidase (rHuPH20)
  Arms: Commercial Hylenex Recombinant (Formulation 1)
Drug: Precommercial Hylenex recombinant (hyaluronidase human injection)
  Other Names: Formulation 2; Hylenex; rHuPH20
  Arms: Precommercial Hylenex Recombinant (Formulation 2)
Drug: Insulin lispro
  Other Names: Humalog; Lispro
Drug: Insulin aspart
  Other Names: Novolog; Aspart
Drug: Insulin glulisine
  Other Names: Apidra; Glulisine

SUMMARY:
The primary objectives of this study are to compare the difference in glycosylated hemoglobin (HbA1c) from baseline to Month 6 using Hylenex recombinant preadministration in continuous subcutaneous insulin infusion (CSII) versus standard CSII and to evaluate the safety of Hylenex recombinant preadministration, including local tolerability, adverse events, and hypo- and hyperglycemia rates.

DETAILED DESCRIPTION:
This Phase 4 study is designed to demonstrate noninferiority of pretreatment with Hylenex recombinant in the CSII setting to rapid-acting analog insulin alone with respect to glycemic control as assessed by changes in HbA1c in participants with Type 1 diabetes mellitus.

Total duration of study treatment is 24 months. However, according to the study design, the primary outcome measure is to be assessed at 6 months and an interim analysis is to be completed at 6 months for the secondary outcome measures and adverse events. Therefore, data reported in this clinical trials record is for the 6-month interim analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of age 18 years or older with a history of T1DM for at least 12 months
2. Glycosylated hemoglobin (HbA1c) 6.5% to 9.5% (inclusive) based on central laboratory results
3. Fasting C-peptide <0.6 nanograms per milliliter (ng/mL)
4. Current use of an insulin pump compatible with available tubing for Hylenex recombinant infusion and use of an infusion set compatible with the tubing available or willingness to switch to an infusion set compatible with tubing available for infusion of Hylenex recombinant
5. Current treatment at the time of screening with insulin <300 units per day (U/day)
6. Participants who routinely use continuous glucose monitoring (CGM) (defined as average CGM use 5 or more days per week over the preceding 3 months) and those who do not routinely used CGM are both eligible for inclusion in the study. Intermittent use of CGM is also acceptable but will not be a criterion use for stratified randomization.
7. Participants should be in good general health based on medical history and physical examination, without medical conditions that might prevent the completion of study drug infusions and assessments required in this protocol.

Exclusion Criteria:

1. Type 2 diabetes
2. Known or suspected allergy to any component of any of the study drugs in this study
3. Severe proliferative retinopathy or maculopathy, and/or gastroparesis, and/or severe neuropathy, in particular autonomic neuropathy, of such severity as to impede the participant's ability to comply with protocol procedures, as judged by the Investigator
4. History of transmural myocardial infarction, congestive heart failure and uncontrolled hypertension (diastolic blood pressure [BP] consistently >100 millimeters of mercury [mmHg]) are exclusionary
5. As judged by the Investigator, clinically significant active disease of the gastrointestinal, cardiovascular (including history of stroke, history of arrhythmia, or conduction delays on electrocardiogram [ECG]), hepatic, neurological, renal, genitourinary, pulmonary, or hematological systems of such severity as to impede the participant's ability to comply with protocol procedures
6. History of any illness or disease that in the opinion of the Investigator might confound the results of the study or pose additional risk in administering the study drugs to the participant
7. As judged by the Investigator, clinically significant findings in routine laboratory data at screening
8. Use of drugs that may interfere with the interpretation of study results or are known to cause clinically relevant interference with hyaluronidase action, insulin action, glucose utilization, or recovery from hypoglycemia (including systemic pharmacologic corticosteroid). Use of pramlintide or a glucagon-like peptide [GLP]-1 receptor agonist is not exclusionary but participants using these agents will be subjected to stratified randomization. Use of aspirin (acetylsalicylic acid [ASA]) up to 325 milligrams (mg)/day is not exclusionary but should be noted for analysis.
9. Hypoglycemic unawareness of such severity as to impede the participant's ability to comply with protocol procedures, as judged by the Investigator.
10. Current addiction to alcohol or substance abuse as determined by the Investigator.
11. Pregnancy, breast-feeding, the intention of becoming pregnant, or not using adequate contraceptive measures (adequate contraceptive measures consist of sterilization, intra-uterine device [IUD], oral or injectable contraceptives, and/or barrier methods). Abstinence alone is not considered an adequate contraceptive measure for the purposes of this study.
12. Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Muchmore, MD, Study Director — Halozyme Therapeutics
Locations (38):
- United States (38):
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Concord, California
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Encino, California
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Escondido, California
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Greenbrae, California
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, La Jolla, California
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, San Mateo, California
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Aurora, Colorado
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Hollywood, Florida
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Miami, Florida
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Roswell, Georgia
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Wichita, Kansas
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Hyattsville, Maryland
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Rockville, Maryland
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Detroit, Michigan
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Butte, Montana
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Henderson, Nevada
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, New Hyde Park, New York
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Durham, North Carolina
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Morehead City, North Carolina
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Portland, Oregon
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Bartlett, Tennessee
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Austin, Texas
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Dallas, Texas
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Round Rock, Texas
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, San Antonio, Texas
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Olympia, Washington
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Renton, Washington
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Seattle, Washington
  - For additional information regarding investigative sites for this trial, call (858) 794-8889 8 AM to 5 PM Mon-Fri Pacific Standard Time, Madison, Wisconsin

REFERENCES:
- See also: Related Info — http://www.halozyme.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Commercial Hylenex Recombinant (Formulation 1): Hylenex Formulation 1: For 12 months, participants received their regular treatment of rapid-acting continuous subcutaneous insulin infusion (CSII) (for example, insulin lispro, insulin aspart, and insulin glulisine). Additionally, during this 12-month treatment period, the participants received a pretreatment dose of the commercial form of Hylenex recombinant, delivered at 150 units (U) through their insulin infusion cannula each time they changed infusion sets (every 2 to 3 days).
- Precommercial Hylenex Recombinant (Formulation 2): Hylenex Formulation 2: For 12 months, participants received their regular treatment of rapid-acting CSII (for example, insulin lispro, insulin aspart, and insulin glulisine). Additionally, during this 12-month treatment period, the participants received a pretreatment dose of the precommercial form of Hylenex recombinant, delivered at 150 U through their insulin infusion cannula each time they changed infusion sets (every 2 to 3 days).
- Standard Rapid-Acting Insulin CSII: Participants received their regular treatment of rapid-acting CSII (for example, insulin lispro, insulin aspart, and insulin glulisine) for 12 months.
Period: Overall Study
Arm/Group | Commercial Hylenex Recombinant (Formulation 1) | Precommercial Hylenex Recombinant (Formulation 2) | Standard Rapid-Acting Insulin CSII
Started | 227 | 115 | 114 (One participant was randomized and withdrew consent before start of study treatment.)
Received at Least 1 Dose of Study Drug | 227 | 115 | 113
Completed Month 6 | 194 | 106 | 103
Completed | 181 | 95 | 98
Not Completed | 46 | 20 | 16
Not completed — Adverse Event | 6 | 2 | 0
Not completed — Lost to Follow-up | 6 | 2 | 2
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 29 | 10 | 11
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Non Compliance | 1 | 0 | 0
Not completed — Death | 1 | 0 | 1
Not completed — Other | 1 | 4 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Commercial Hylenex Recombinant (Formulation 1): Hylenex Formulation 1: For 12 months, participants received their regular treatment of rapid-acting continuous CSII (for example, insulin lispro, insulin aspart, and insulin glulisine). Additionally, during this 12-month treatment period, the participants received a pretreatment dose of the commercial form of Hylenex recombinant, delivered at 150 U through their insulin infusion cannula each time they changed infusion sets (every 2 to 3 days).
- Total: Total of all reporting groups
Arm/Group | Commercial Hylenex Recombinant (Formulation 1) | Precommercial Hylenex Recombinant (Formulation 2) | Standard Rapid-Acting Insulin CSII | Total
Number analyzed (Participants) | 227 | 115 | 113 | 455
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (12.90) | 45.9 (13.14) | 49.7 (14.73) | 47.6 (13.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 53 | 64 | 239
  Male | 105 | 62 | 49 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 5 | 22
  Not Hispanic or Latino | 217 | 108 | 108 | 433
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 3 | 0 | 2 | 5
  Black or African American | 8 | 3 | 2 | 13
  White | 216 | 112 | 107 | 435
  Asian Indian | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 227 | 115 | 113 | 455

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 6 Months in Glycosylated Hemoglobin (HbA1c)
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; 6 Months
Population: Participants who received at least one dose of study drug and had evaluable HbA1c data. Comparisons were made by pooling all of the rHuPH20 pretreatment participants (including both Formulations 1 and 2) and comparing against the standard CSII treatment arm. Formulation 1 versus Formulation 2 was compared as a supportive analysis.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Groups:
- Hylenex Recombinant: For 6 months, participants received their regular treatment of rapid-acting Continuous Subcutaneous Insulin Infusion (CSII) (for example, insulin lispro, insulin aspart, and insulin glulisine). Additionally, during this 6-month treatment period, the participants received a pretreatment dose of Hylenex recombinant (either Formulation 1 or Formulation 2), delivered at 150 U through their insulin infusion cannula each time they changed infusion sets (every 2 to 3 days).
- Standard Rapid-Acting Insulin CSII: Participants received their regular treatment of rapid-acting insulin CSII (for example, insulin lispro, insulin aspart, and insulin glulisine) for 6 months.
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 296 | 103
percentage of HbA1c | -0.14 (0.521) | -0.18 (0.687)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Sample size calculated based on approximately 400 participants (Pt) being enrolled. No more than 10% dropout rate at 6 months allowed at least 270 Hylenex and 90 standard CSII Pt to reach primary metabolic endpoint evaluation. Assuming HbA1c standard deviation of 0.7% and population difference of 0% between treatments, Pt reaching primary efficacy endpoint would provide >90% power to demonstrate HbA1c noninferiority at margin of 0.4% using confidence bound from 2-tailed 95% confidence interval; Test type: Non-Inferiority or Equivalence — If the upper bound of the 95% CI for the treatment difference ≤0.40, it is concluded that Hylenex recombinant preadministration is noninferior to standard CSII; p = 0.4516, ANOVA; Analysis of variance (ANOVA) with treatment (Hylenex, standard rapid-acting insulin CSII) as a fixed effect; least squares mean treatment difference = 0.05, 95% CI 2-sided [-0.08 to 0.18] — Hylenex minus Standard CSII

2. Primary Outcome: Change From Baseline to 12 Months in HbA1c
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; 12 Months
Population: Intent-to-Treat (ITT) Population: all randomized participants (par.). Comparisons were made by pooling all rHuPH20 pretreatment par. (including both Formulations 1 and 2) and comparing against the standard CSII treatment arm. Formulation 1 versus Formulation 2 was compared as a supportive analysis. Only par. with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Groups:
- Hylenex Recombinant: For 12 months, participants received their regular treatment of rapid-acting CSII (for example, insulin lispro, insulin aspart, and insulin glulisine). Additionally, during this 12-month treatment period, the participants received a pretreatment dose of Hylenex recombinant (either Formulation 1 or Formulation 2), delivered at 150 U through their insulin infusion cannula each time they changed infusion sets (every 2 to 3 days).
- Standard Rapid-Acting Insulin CSII: Participants received their regular treatment of rapid-acting insulin CSII (for example, insulin lispro, insulin aspart, and insulin glulisine) for 12 months.
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 268 | 95
percentage of HbA1c | -0.13 (0.590) | -0.26 (0.718)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Sample size calculated based on approximately 400 Pt being enrolled. No more than 10% dropout rate at 6 months allowed at least 270 Hylenex and 90 standard CSII Pt to reach primary metabolic endpoint evaluation. Assuming HbA1c standard deviation of 0.7% and population difference of 0% between treatments, Pt reaching primary efficacy endpoint would provide >90% power to demonstrate HbA1c noninferiority at margin of 0.4% using confidence bound from 2-tailed 95% confidence interval; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0711, ANOVA; ANOVA with treatment (Hylenex, standard rapid-acting insulin CSII) as a fixed effect; least squares mean treatment difference = 0.14, 95% CI 2-sided [-0.01 to 0.28] — Hylenex minus Standard CSII

3. Secondary Outcome: Rates of Hypoglycemia Events (HE) to Month 6
Description: Overall rates of hypoglycemia (defined as blood glucose ≤70 milligrams per deciliter [mg/dL] and <56 mg/dL) were based on measurements after 1 month up to 6 months. A severe HE was classified as an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. A nocturnal HE was classified as an event with a blood glucose of ≤70 mg/dL with start time between 2300 and 0600, inclusive. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module. Comparisons were made by pooling all of the rHuPH20 pretreatment participants (including both Formulations 1 and 2) and comparing against the standard CSII treatment arm. Formulation 1 versus Formulation 2 was compared as a supportive analysis.
Time Frame: After Month 1 up to Month 6
Population: Primary Self-Monitoring of Blood Glucose (SMBG) Analysis Population: all randomized participants who received study treatment and had SMBG data up to Month 6. Only participants with available data were analyzed. The "Number Analyzed" reflects the number of participants with at least one event.
Measure: Number; unit: events per participant per month
Groups:
- Hylenex Recombinant: For 6 months, participants received their regular treatment of rapid-acting CSII (for example, insulin lispro, insulin aspart, and insulin glulisine). Additionally, during this 6-month treatment period, the participants received a pretreatment dose of Hylenex recombinant (either Formulation 1 or Formulation 2), delivered at 150 U through their insulin infusion cannula each time they changed infusion sets (every 2 to 3 days).
Arm/Group | Hylenex Recombinant | Standard Rapid-acting Insulin CSII
Number analyzed (Participants) | 184 | 63
events per participant per month
  <56 mg/dL: number analyzed (Participants) | 167 | 60
  <56 mg/dL | 2.9103 | 4.1970
  ≤70 mg/dL | 11.6219 | 14.7112
  Nocturnal HEs: number analyzed (Participants) | 174 | 58
  Nocturnal HEs | 1.6224 | 2.0727
  Severe HEs: number analyzed (Participants) | 5 | 4
  Severe HEs | 0.0055 | 0.0160
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.0105, negative binomial model — SMBG <56 mg/dL; rate ratio = 0.69 — Hylenex/Standard CSII
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.0130, negative binomial model — SMBG <=70 mg/dL; rate ratio = 0.79 — Hylenex/Standard CSII
Statistical Analysis 3: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.0511, negative binomial model — Nocturnal HEs; rate ratio = 0.78 — Hylenex/Standard CSII
Statistical Analysis 4: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.1176, negative binomial model — Severe HEs; rate ratio = 0.34 — Hylenex/Standard CSII

4. Secondary Outcome: Rates of HEs to Month 12
Description: Overall rates of hypoglycemia (defined as blood glucose ≤70 milligrams per deciliter [mg/dL] and <56 mg/dL) were based on measurements after 1 month up to 12 months. A severe HE was classified as an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. A nocturnal HE was classified as an event with a blood glucose of ≤70 mg/dL with start time between 2300 and 0600, inclusive. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module. Comparisons were made by pooling all of the rHuPH20 pretreatment participants (including both Formulations 1 and 2) and comparing against the standard CSII treatment arm. Formulation 1 versus Formulation 2 was compared as a supportive analysis.
Time Frame: After Month 1 up to Month 12
Population: ITT Population. Only participants with available data were analyzed. The "Number Analyzed" reflects the number of participants with at least one event.
Measure: Number; unit: events per participant per month
Arm/Group | Hylenex Recombinant | Standard Rapid-acting Insulin CSII
Number analyzed (Participants) | 342 | 114
events per participant per month
  <56 mg/dL: number analyzed (Participants) | 320 | 106
  <56 mg/dL | 2.6792 | 3.3022
  ≤70 mg/dL: number analyzed (Participants) | 339 | 112
  ≤70 mg/dL | 11.3803 | 12.3591
  Nocturnal HEs: number analyzed (Participants) | 319 | 107
  Nocturnal HEs | 1.6754 | 1.9203
  Severe HEs: number analyzed (Participants) | 23 | 7
  Severe HEs | 0.0091 | 0.0085
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.0456, negative binomial model — SMBG <56 mg/dL; rate ratio = 0.81 — Hylenex/Standard CSII
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.2322, negative binomial model — SMBG <=70 mg/dL; rate ratio = 0.92 — Hylenex/Standard CSII
Statistical Analysis 3: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.1365, negative binomial model — Nocturnal HEs; rate ratio = 0.87 — Hylenex/Standard CSII
Statistical Analysis 4: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.8909, negative binomial model — Severe HEs; rate ratio = 1.07 — Hylenex/Standard CSII

5. Secondary Outcome: Rates of Hyperglycemia Events to Month 6
Description: Overall rates of hyperglycemia (defined as blood glucose >240 mg/dL and >300 mg/dL) were based on measurements after 1 month up to 6 months. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module. Comparisons were made by pooling all of the rHuPH20 pretreatment participants (including both Formulations 1 and 2) and comparing against the standard CSII treatment arm. Formulation 1 versus Formulation 2 was compared as a supportive analysis.
Time Frame: After Month 1 up to Month 6
Population: Primary SMBG Analysis Population. Only participants with available data were analyzed. The "Number Analyzed" reflects the number of participants with at least one event.
Measure: Number; unit: events per participant per month
Arm/Group | Hylenex Recombinant | Standard Rapid-acting Insulin CSII
Number analyzed (Participants) | 298 | 103
events per participant per month
  >240 mg/dL: number analyzed (Participants) | 296 | 103
  >240 mg/dL | 18.0422 | 18.4696
  >300 mg/dL: number analyzed (Participants) | 293 | 102
  >300 mg/dL | 6.4768 | 6.8155
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.7292, negative binomial model — SMBG >240 mg/dL; rate ratio = 0.98 — Hylenex/Standard CSII
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.5895, negative binomial model — SMBG >300 mg/dL; rate ratio = 0.95 — Hylenex/Standard CSII

6. Secondary Outcome: Rates of Hyperglycemia Events to Month 12
Description: Overall rates of hyperglycemia (defined as blood glucose >240 mg/dL and >300 mg/dL) were based on measurements after 1 month up to 12 months. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module. Comparisons were made by pooling all of the rHuPH20 pretreatment participants (including both Formulations 1 and 2) and comparing against the standard CSII treatment arm. Formulation 1 versus Formulation 2 was compared as a supportive analysis.
Time Frame: After Month 1 up to Month 12
Population: as for outcome 4
Measure: Number; unit: events per participant per month
Arm/Group | Hylenex Recombinant | Standard Rapid-acting Insulin CSII
Number analyzed (Participants) | 342 | 114
events per participant per month
  >240 mg/dL: number analyzed (Participants) | 338 | 113
  >240 mg/dL | 18.9784 | 18.2785
  >300 mg/dL: number analyzed (Participants) | 336 | 110
  >300 mg/dL | 7.1138 | 6.8900
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.5414, negative binomial model — SMBG >240 mg/dL; rate ratio = 1.04 — Hylenex/Standard CSII
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.7110, negative binomial model — SMBG >300 mg/dL; rate ratio = 1.03 — Hylenex/Standard CSII

7. Secondary Outcome: Mean Glucose Excursions at 6 Months
Description: A 4-hour postprandial glucose excursion was measured for 3 meals after 1 month up to 6 months. For each of the 3 meals, the mealtime (breakfast, lunch, and dinner) excursions were calculated as the post-meal glucose value minus the pre-meal (for measurements taken within 15 minutes before a meal). The average of all excursions is presented. Least Squares (LS) means were calculated from ANOVA with treatment (Hylenex, standard rapid-acting insulin CSII) as a fixed effect. Comparisons were made by pooling all of the rHuPH20 pretreatment participants (including both Formulations 1 and 2) and comparing against the standard CSII treatment arm. Formulation 1 versus Formulation 2 was compared as a supportive analysis.
Time Frame: After Month 1 up to Month 6
Population: Primary SMBG Analysis Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Hylenex Recombinant | Standard Rapid-acting Insulin CSII
Number analyzed (Participants) | 184 | 63
milligrams per deciliter (mg/dL)
  Breakfast: number analyzed (Participants) | 180 | 61
  Breakfast | 17.3 (2.77) | 20.7 (4.76)
  Lunch: number analyzed (Participants) | 182 | 62
  Lunch | 22.2 (2.67) | 17.9 (4.58)
  Dinner: number analyzed (Participants) | 181 | 62
  Dinner | 12.6 (2.45) | 12.5 (4.18)
  Overall: number analyzed (Participants) | 182 | 62
  Overall | 17.1 (1.70) | 16.9 (2.91)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.5394, ANOVA — Breakfast; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -3.4, 95% CI 2-sided [-14.2 to 7.5] — Hylenex minus Standard CSII
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.4151, ANOVA — Lunch; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 4.3, 95% CI 2-sided [-6.1 to 14.8] — Hylenex minus Standard CSII
Statistical Analysis 3: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.9930, ANOVA — Dinner; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.0, 95% CI 2-sided [-9.5 to 9.6] — Hylenex minus Standard CSII
Statistical Analysis 4: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.9410, ANOVA — Overall; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.2, 95% CI 2-sided [-6.4 to 6.9] — Hylenex minus Standard CSII

8. Secondary Outcome: Mean Glucose Excursions at 12 Months
Description: A 4-hour postprandial glucose excursion was measured for 3 meals after 1 month up to 12 months. For each of the 3 meals, the mealtime (breakfast, lunch, and dinner) excursions were calculated as the post-meal glucose value minus the pre-meal (for measurements taken within 15 minutes before a meal). The average of all excursions is presented. LS means were calculated from ANOVA with treatment (Hylenex, standard rapid-acting insulin CSII) as a fixed effect. Comparisons were made by pooling all of the rHuPH20 pretreatment participants (including both Formulations 1 and 2) and comparing against the standard CSII treatment arm. Formulation 1 versus Formulation 2 was compared as a supportive analysis.
Time Frame: After Month 1 up to Month 12
Population: ITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Hylenex Recombinant | Standard Rapid-acting Insulin CSII
Number analyzed (Participants) | 200 | 63
milligrams per deciliter (mg/dL)
  Breakfast: number analyzed (Participants) | 197 | 62
  Breakfast | 20.1 (2.36) | 24.9 (4.21)
  Lunch: number analyzed (Participants) | 198 | 62
  Lunch | 22.4 (2.17) | 21.0 (3.89)
  Dinner: number analyzed (Participants) | 198 | 63
  Dinner | 12.7 (2.08) | 13.8 (3.69)
  Overall: number analyzed (Participants) | 199 | 63
  Overall | 17.1 (1.49) | 19.7 (2.65)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.3239, ANOVA — Breakfast; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -4.8, 95% CI 2-sided [-14.3 to 4.7] — Hylenex minus Standard CSII
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.7540, ANOVA — Lunch; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 1.4, 95% CI 2-sided [-7.4 to 10.2] — Hylenex minus Standard CSII
Statistical Analysis 3: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.7904, ANOVA — Dinner; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -1.1, 95% CI 2-sided [-9.5 to 7.2] — Hylenex minus Standard CSII
Statistical Analysis 4: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.4016, ANOVA — Overall; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -2.6, 95% CI 2-sided [-8.5 to 3.4] — Hylenex minus Standard CSII

9. Secondary Outcome: Standard Deviation of Self-Monitoring Blood Glucose Values at 6 Months
Description: Standard deviation of self-monitoring blood glucose values was calculated based on measurements taken within 15 minutes before a meal, 1 month and up to 6 months after study drug administration. LS means were calculated from ANOVA with treatment (Hylenex, standard rapid-acting insulin CSII) as a fixed effect. Comparisons were made by pooling all of the rHuPH20 pretreatment participants (including both Formulations 1 and 2) and comparing against the standard CSII treatment arm. Formulation 1 versus Formulation 2 was compared as a supportive analysis.
Time Frame: After Month 1 up to Month 6
Population: Primary SMBG Analysis Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Hylenex Recombinant | Standard Rapid-acting Insulin CSII
Number analyzed (Participants) | 184 | 63
mg/dL | 70.9 (1.09) | 72.2 (1.86)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.5260, ANOVA; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -1.4, 95% CI 2-sided [-5.6 to 2.9] — Hylenex minus Standard CSII

10. Secondary Outcome: Standard Deviation of Self-Monitoring Blood Glucose Values at 12 Months
Description: Standard deviation of self-monitoring blood glucose values was calculated based on measurements taken within 15 minutes before a meal, 1 month and up to 12 months after study drug administration. LS means were calculated from ANOVA with treatment (Hylenex, standard rapid-acting insulin CSII) as a fixed effect. Comparisons were made by pooling all of the rHuPH20 pretreatment participants (including both Formulations 1 and 2) and comparing against the standard CSII treatment arm. Formulation 1 versus Formulation 2 was compared as a supportive analysis.
Time Frame: After Month 1 up to Month 12
Population: ITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Hylenex Recombinant | Standard Rapid-acting Insulin CSII
Number analyzed (Participants) | 200 | 63
mg/dL | 72.9 (1.04) | 72.4 (1.85)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.8049, ANOVA; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.5, 95% CI 2-sided [-3.7 to 4.7] — Hylenex minus Standard CSII

11. Secondary Outcome: Number of Participants Achieving HbA1c <7.0% and HbA1c ≤6.5% at Month 12
Description: The number of participants achieving HbA1c goals of <7% and ≤6.5% was calculated.
Time Frame: Month 12
Population: ITT Population. Only participants with available data were analyzed. Comparisons were made by pooling all of the rHuPH20 pretreatment participants (including both Formulations 1 and 2) and comparing against the standard CSII treatment arm. Formulation 1 versus Formulation 2 was compared as a supportive analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 268 | 95
Participants
  HbA1c <7.0% | 61 | 21
  HbA1c ≤6.5% | 18 | 6
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.8955, Chi-squared — HbA1c <7.0%
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.8926, Chi-squared — HbA1c ≤6.5%

12. Secondary Outcome: Change From Baseline in Body Weight to Month 12
Description: Baseline is defined as the last measurement prior to randomization.
Time Frame: Baseline; Week 2; Months 1, 2, 3, 4, 6, 9, and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 342 | 114
kilograms
  Week 2: number analyzed (Participants) | 334 | 111
  Week 2 | -0.10 (1.272) | 0.19 (1.257)
  Month 1: number analyzed (Participants) | 327 | 111
  Month 1 | -0.11 (1.583) | 0.20 (1.696)
  Month 2: number analyzed (Participants) | 320 | 107
  Month 2 | -0.03 (2.002) | 0.48 (1.672)
  Month 3: number analyzed (Participants) | 315 | 105
  Month 3 | 0.16 (2.562) | 0.37 (1.858)
  Month 4: number analyzed (Participants) | 308 | 105
  Month 4 | 0.04 (2.680) | 0.37 (2.230)
  Month 6: number analyzed (Participants) | 297 | 102
  Month 6 | 0.60 (3.035) | 0.83 (2.287)
  Month 9: number analyzed (Participants) | 281 | 102
  Month 9 | 0.91 (3.355) | 0.92 (3.033)
  Month 12: number analyzed (Participants) | 276 | 98
  Month 12 | 0.61 (3.796) | 0.48 (4.078)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.7735, ANOVA; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.13, 95% CI 2-sided [-0.76 to 1.03] — Hylenex minus Standard CSII

13. Secondary Outcome: Average of Daily Insulin Doses (Bolus, Basal, and Total)
Description: The daily bolus insulin dose is calculated as the daily prandial (occurring before a meal) insulin dose plus the daily corrective insulin dose. Cumulative basal dosage is to generally be within 40% to 60% of the total daily dose.
Time Frame: from Randomization up to Month 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: International units
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 327 | 111
International units
  Daily bolus dose | 21.9 (0.78) | 22.9 (1.33)
  Daily basal dose | 28.0 (0.73) | 25.7 (1.26)
  Daily total dose | 49.9 (1.32) | 48.5 (2.27)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.4948, ANOVA — Daily bolus dose; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -1.1, 95% CI 2-sided [-4.1 to 2.0] — Hylenex minus Standard CSII
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.1099, ANOVA — Daily basal dose; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 2.3, 95% CI 2-sided [-0.5 to 5.2] — Hylenex minus Standard CSII
Statistical Analysis 3: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.5830, ANOVA — Daily total dose; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 1.4, 95% CI 2-sided [-3.7 to 6.6] — Hylenex minus Standard CSII

14. Secondary Outcome: Average Carbohydrate Factor (CarbF) Values
Description: CarbF is calculated as 2.6 * weight (pounds) / total daily dose of insulin (grams per unit).
Time Frame: Month 1 to Month 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: grams per unit
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 304 | 100
grams per unit | 11.1 (0.26) | 11.0 (0.46)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.8778, ANOVA; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.1, 95% CI 2-sided [-1.0 to 1.1] — Hylenex minus Standard CSII

15. Secondary Outcome: Average Correction Factor (CorrF) Values
Description: CorrF is calculated as 1960 / total daily dose of insulin (milligrams/[deciliter*unit]).
Time Frame: Month 1 to Month 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: milligrams/(deciliter*unit)
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 299 | 101
milligrams/(deciliter*unit) | 43.2 (1.06) | 45.3 (1.83)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.3233, ANOVA; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -2.1, 95% CI 2-sided [-6.3 to 2.1] — Hylenex minus Standard CSII

16. Secondary Outcome: Average of Bolus Times Relative to Meal Times
Description: The average meal bolus timing relative to meal time is defined as the minutes between the start time of a meal bolus and the start time of a meal.
Time Frame: Month 1 to Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 342 | 114
minutes
  Breakfast: number analyzed (Participants) | 302 | 101
  Breakfast | -2.3 (8.17) | -3.9 (7.83)
  Lunch: number analyzed (Participants) | 303 | 101
  Lunch | -1.8 (6.75) | -1.6 (8.61)
  Dinner: number analyzed (Participants) | 303 | 101
  Dinner | -1.7 (7.48) | -1.7 (9.19)
  Overall: number analyzed (Participants) | 303 | 101
  Overall | -1.9 (6.51) | -2.4 (7.86)

17. Secondary Outcome: Average Glucose, Median Glucose, and Average Daily Standard Deviation
Description: For each participant, the following continuous glucose monitoring (CGM) parameters were calculated using CGM values recorded after Randomization up to Month 12: average glucose, median glucose, and average daily standard deviation.
Time Frame: Randomization to Month 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: milliliters per deciliter
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 80 | 30
milliliters per deciliter
  Average glucose | 152.9 (1.79) | 151.9 (2.93)
  Median glucose | 145.2 (1.80) | 143.4 (2.94)
  Average daily standard deviation | 48.9 (0.85) | 49.7 (1.39)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.7708, ANOVA — Average glucose; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 1.0, 95% CI 2-sided [-5.8 to 7.8] — Hylenex minus Standard CSII
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.6058, ANOVA — Median glucose; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 1.8, 95% CI 2-sided [-5.0 to 8.6] — Hylenex minus Standard CSII
Statistical Analysis 3: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.6571, ANOVA — Average daily standard deviation; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -0.7, 95% CI 2-sided [-4.0 to 2.5] — Hylenex minus Standard CSII

18. Secondary Outcome: Time Per Day <56 Milligrams Per Deciliter (mg/dL), ≤70 mg/dL, >70 mg/dL, <140 mg/dL, ≥140 mg/dL, Outside of 71 to 180 mg/dL, and Outside of 71 to 139 mg/dL
Description: For each participant, the following CGM parameters were calculated using CGM values recorded after Randomization up to Month 12: time per day spent in the pre-defined glucose classes.
Time Frame: Randomization to Month 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 80 | 30
minutes
  Time per day <56 mg/dL | 18.1 (2.40) | 20.3 (3.91)
  Time per day ≤70 mg/dL | 63.0 (5.37) | 68.5 (8.77)
  Time per day >70 mg/dL | 1358.8 (5.62) | 1351.9 (9.18)
  Time per day <140 mg/dL | 660.3 (16.99) | 683.7 (27.74)
  Time per day ≥140 mg/dL | 756.4 (17.02) | 732.5 (27.80)
  Time per day outside of 71 to 180 mg/dL | 464.4 (15.02) | 461.7 (24.54)
  Time per day outside of 71 to139 mg/dL | 819.4 (14.74) | 801.0 (24.07)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.6252, ANOVA — Time per day <56 mg/dL; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -2.2, 95% CI 2-sided [-11.3 to 6.9] — Hylenex minus Standard CSII
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.5929, ANOVA — Time per day ≤70 mg/dL; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -5.5, 95% CI 2-sided [-25.9 to 14.9] — Hylenex minus Standard CSII
Statistical Analysis 3: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.5207, ANOVA — Time per day >70 mg/dL; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 6.9, 95% CI 2-sided [-14.4 to 28.3] — Hylenex minus Standard CSII
Statistical Analysis 4: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.4754, ANOVA — Time per day <140 mg/dL; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -23.3, 95% CI 2-sided [-87.8 to 41.2] — Hylenex minus Standard CSII
Statistical Analysis 5: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.4644, ANOVA — Time per day ≥140 mg/dL; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 23.9, 95% CI 2-sided [-40.7 to 88.6] — Hylenex minus Standard CSII
Statistical Analysis 6: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.9232, ANOVA — Time per day outside of 71 to 180 mg/dL; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 2.8, 95% CI 2-sided [-54.2 to 59.8] — Hylenex minus Standard CSII
Statistical Analysis 7: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.5151, ANOVA — Time per day outside of 71 to 139 mg/dL; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 18.4, 95% CI 2-sided [-37.5 to 74.4] — Hylenex minus Standard CSII

19. Secondary Outcome: Area Per Day <56 mg/dL, ≤70 mg/dL, ≥140 mg/dL, Outside of 71 to 180 mg/dL, and Outside of 71 to 139 mg/dL
Description: For each participant, the following continuous glucose monitoring (CGM) parameters were calculated using CGM values recorded after Randomization up to Month 12: area per day spent in the pre-defined glucose classes. The area per day for a specific glucose concentration range (e.g., <56 mg/dL) is the sum of the area under the curve with glucose concentration falling in the specific glucose concentration range (e.g., <56 mg/dL). For example, if the glucose stays constant at 50 mg/dL for the whole day (1,440 minutes), the area per day for glucose < 56 mg/dL equals: 50*1440 = 72,000 mg*minutes/dL.
Time Frame: Randomization to Month 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: mg*minutes/deciliter
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 80 | 30
mg*minutes/deciliter
  Area per day <56 mg/dL | 129.7 (21.71) | 163.2 (35.45)
  Area per day ≤70 mg/dL | 687.0 (77.58) | 771.7 (126.69)
  Area per day ≥140 mg/dL | 42660.2 (1874.62) | 42317.2 (3061.24)
  Area per day outside of 71 to 180 mg/dL | 20033.8 (1232.60) | 20411.2 (2012.83)
  Area per day outside of 71 to 139 mg/dL | 43347.2 (1857.54) | 43089.0 (3033.35)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.4216, ANOVA — Area per day <56 mg/dL; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -33.5, 95% CI 2-sided [-115.9 to 48.9] — Hylenex minus Standard CSII
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.5697, ANOVA — Area per day ≤70 mg/dL; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -84.7, 95% CI 2-sided [-379.2 to 209.8] — Hylenex minus Standard CSII
Statistical Analysis 3: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.9241, ANOVA — Area per day ≥140 mg/dL; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 342.9, 95% CI 2-sided [-6772.3 to 7458.2] — Hylenex minus Standard CSII
Statistical Analysis 4: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.9232, ANOVA — Area per day outside of 71 to 180 mg/dL; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 2.8, 95% CI 2-sided [-54.2 to 59.8] — Hylenex minus Standard CSII
Statistical Analysis 5: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.9423, ANOVA — Area per day outside of 71 to 139 mg/dL; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; Mean Difference (Final Values) = 258.2, 95% CI 2-sided [-6792.2 to 7308.7] — Least squares mean treatment difference (Hylenex minus Standard CSII)

20. Secondary Outcome: Change From Baseline in Weighted Impact ADDQoL Values at Month 12
Description: The Audit of Diabetes Dependent Quality of Life (ADDQoL) is a validated, diabetes-specific questionnaire to evaluate the participant's assessment of quality of life (QoL). Participants rated the impact of diabetes on 19 applicable domains on a scale from -3 (maximum negative impact) to +3 (maximum positive impact) and then rated the importance of those domains for their QoL on a scale from 3 (very important) to 0 (not at all important). Impact ratings were multiplied by the corresponding importance ratings to provide a weighted-impact score for each domain from -9 (maximum negative impact) to +9 (maximum positive impact).
Time Frame: Baseline; Month 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 342 | 114
score on a scale
  Leisure activities: number analyzed (Participants) | 264 | 94
  Leisure activities | -0.2 (0.14) | 0.0 (0.24)
  Work life: number analyzed (Participants) | 203 | 63
  Work life | -0.1 (0.15) | 0.0 (0.27)
  Local or long distance travel: number analyzed (Participants) | 264 | 94
  Local or long distance travel | -0.4 (0.15) | -0.2 (0.25)
  Vacations: number analyzed (Participants) | 255 | 86
  Vacations | 0.0 (0.15) | 0.2 (0.25)
  Do physically: number analyzed (Participants) | 259 | 93
  Do physically | -0.1 (0.14) | -0.2 (0.23)
  Family life: number analyzed (Participants) | 257 | 94
  Family life | 0.2 (0.14) | 0.1 (0.23)
  Friendships and social life: number analyzed (Participants) | 261 | 94
  Friendships and social life | 0.3 (0.13) | 0.1 (0.22)
  Close personal relationship: number analyzed (Participants) | 246 | 86
  Close personal relationship | 0.1 (0.16) | 0.1 (0.27)
  Sex life: number analyzed (Participants) | 250 | 83
  Sex life | 0.0 (0.14) | -0.3 (0.24)
  Physical appearance: number analyzed (Participants) | 265 | 93
  Physical appearance | 0.1 (0.11) | -0.2 (0.19)
  Self-confidence: number analyzed (Participants) | 267 | 94
  Self-confidence | 0.0 (0.12) | -0.1 (0.21)
  Motivation: number analyzed (Participants) | 263 | 94
  Motivation | 0.0 (0.14) | 0.3 (0.24)
  The way people in general react: number analyzed (Participants) | 263 | 95
  The way people in general react | 0.2 (0.10) | -0.1 (0.17)
  Feelings about the future: number analyzed (Participants) | 264 | 95
  Feelings about the future | -0.1 (0.16) | 0.3 (0.26)
  Financial situation: number analyzed (Participants) | 264 | 94
  Financial situation | 0.1 (0.14) | 0.0 (0.23)
  Living situation and conditions: number analyzed (Participants) | 264 | 95
  Living situation and conditions | 0.0 (0.13) | -0.1 (0.22)
  Depend on others: number analyzed (Participants) | 264 | 95
  Depend on others | -0.1 (0.17) | 0.4 (0.28)
  Freedom to eat: number analyzed (Participants) | 263 | 94
  Freedom to eat | 0.0 (0.15) | -0.3 (0.25)
  Freedom to drink: number analyzed (Participants) | 267 | 95
  Freedom to drink | -0.2 (0.14) | -0.3 (0.23)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.5246, ANOVA — Leisure activities; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -0.2, 95% CI 2-sided [-0.7 to 0.4] — Hylenex minus Standard CSII
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.6380, ANOVA — Work life; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -0.1, 95% CI 2-sided [-0.8 to 0.5] — Hylenex minus Standard CSII
Statistical Analysis 3: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.5719, ANOVA — Local or long distance travel; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -0.2, 95% CI 2-sided [-0.7 to 0.4] — Hylenex minus Standard CSII
Statistical Analysis 4: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.4052, ANOVA — Vacations; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -0.2, 95% CI 2-sided [-0.8 to 0.3] — Hylenex minus Standard CSII
Statistical Analysis 5: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.7240, ANOVA — Do physically; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.1, 95% CI 2-sided [-0.4 to 0.6] — Hylenex minus Standard CSII
Statistical Analysis 6: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.6876, ANOVA — Family life; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.1, 95% CI 2-sided [-0.4 to 0.6] — Hylenex minus Standard CSII
Statistical Analysis 7: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.6478, ANOVA — Friendships and social life; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.1, 95% CI 2-sided [-0.4 to 0.6] — Hylenex minus Standard CSII
Statistical Analysis 8: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.9744, ANOVA — Close personal relationship; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.0, 95% CI 2-sided [-0.6 to 0.6] — Hylenex minus Standard CSII
Statistical Analysis 9: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.3177, ANOVA — Sex life; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.3, 95% CI 2-sided [-0.3 to 0.8] — Hylenex minus Standard CSII
Statistical Analysis 10: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.2087, ANOVA — Physical appearance; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.3, 95% CI 2-sided [-0.2 to 0.7] — Hylenex minus Standard CSII
Statistical Analysis 11: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.7907, ANOVA — Self-confidence; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.1, 95% CI 2-sided [-0.4 to 0.5] — Hylenex minus Standard CSII
Statistical Analysis 12: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.3444, ANOVA — Motivation; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -0.3, 95% CI 2-sided [-0.8 to 0.3] — Hylenex minus Standard CSII
Statistical Analysis 13: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.2175, ANOVA — The way people in general react; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.2, 95% CI 2-sided [-0.1 to 0.6] — Hylenex minus Standard CSII
Statistical Analysis 14: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.2062, ANOVA — Feelings about the future; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -0.4, 95% CI 2-sided [-1.0 to 0.2] — Hylenex minus Standard CSII
Statistical Analysis 15: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.8762, ANOVA — Financial situation; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.0, 95% CI 2-sided [-0.5 to 0.6] — Hylenex minus Standard CSII
Statistical Analysis 16: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.8900, ANOVA — Living situation and conditions; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.0, 95% CI 2-sided [-0.5 to 0.5] — Hylenex minus Standard CSII
Statistical Analysis 17: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.1367, ANOVA — Depend on others; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = -0.5, 95% CI 2-sided [-1.1 to 0.2] — Hylenex minus Standard CSII
Statistical Analysis 18: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.3144, ANOVA — Freedom to eat; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.3, 95% CI 2-sided [-0.3 to 0.9] — Hylenex minus Standard CSII
Statistical Analysis 19: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.6869, ANOVA — Freedom to drink; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.1, 95% CI 2-sided [-0.4 to 0.6] — Hylenex minus Standard CSII

21. Secondary Outcome: Change From Baseline in Average Weighted Impact ADDQoL Values at Month 12
Description: The ADDQoL is a validated, diabetes-specific questionnaire to evaluate the participant's assessment of QoL. Participants rated the impact of diabetes on 19 applicable domains on a scale from -3 (maximum negative impact) to +3 (maximum positive impact) and then rated the importance of those domains for their QoL on a scale from 3 (very important) to 0 (not at all important). Impact ratings were multiplied by the corresponding importance ratings to provide a weighted-impact score for each domain from -9 (maximum negative impact) to +9 (maximum positive impact). Weighted impact scores were summed and divided by the number of applicable domains to give an overall Average Weighted Impact (AWI) score (higher values represent more positive impact). If there were less than 13 non-missing weighted-impact values, AWI was not to be calculated. Baseline is defined as the last measurement prior to randomization.
Time Frame: Baseline; Month 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 265 | 95
score on a scale | 0.0 (0.07) | 0.0 (0.12)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.9901, ANOVA; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.0, 95% CI 2-sided [-0.3 to 0.3] — Hylenex minus Standard CSII

22. Secondary Outcome: Change From Baseline in DTSQs and DTSQc at Month 12
Description: The Diabetes Treatment Satisfaction Questionnaire-status version (DTSQs) and DTSQ-change version (DTSQc) are validated tools to assess treatment satisfaction and change in treatment satisfaction after therapy changes have occurred. The scale total was computed by adding the 6 items (1, 4, 5, 6, 7, and 8) to produce the Treatment Satisfaction scale total, which has a minimum of 0 and a maximum of 36 on the DTSQs and a minimum of -18 and a maximum of 18 on the DTSQc. Higher scores represent greater satisfaction. If any of the 6 item scores were missing and the numbers of missing scores were less than the number of non-missing scores, the Treatment Satisfaction scale score was to be computed by taking the average of the existing scores and multiplying the average by 6. If there were less than 4 non-missing item scores, the Treatment Satisfaction scale score was not to be calculated. Baseline is defined as the last measurement prior to randomization.
Time Frame: Baseline; Month 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 342 | 114
score on a scale
  DTSQs: number analyzed (Participants) | 261 | 93
  DTSQs | 0.0 (0.32) | 0.0 (0.53)
  DTSQc: number analyzed (Participants) | 267 | 90
  DTSQc | 9.4 (0.40) | 9.4 (0.68)
Statistical Analysis 1: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.9081, ANOVA — DTSQs; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.1, 95% CI 2-sided [-1.1 to 1.3] — Hylenex minus Standard CSII
Statistical Analysis 2: Comparison: Hylenex Recombinant vs Standard Rapid-Acting Insulin CSII; Test type: Non-Inferiority — prespecific non-inferiority margin of 0.4%; p = 0.9840, ANOVA — DTSQc; ANOVA with treatment (Hylenex, Standard CSII) as a fixed effect; least squares mean treatment difference = 0.0, 95% CI 2-sided [-1.5 to 1.6] — Hylenex minus Standard CSII

23. Secondary Outcome: Mean Time to Change Infusion Site
Description: Participants were asked device handling questions to provide information about the impact of the Hylenex administration procedure on everyday life and to investigate perceptions of the overall efficacy and responsiveness of their insulin program.
Time Frame: Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 276 | 97
minutes | 5.7 (4.45) | 4.7 (3.68)

24. Secondary Outcome: Mean Additional Time for Hylenex Pre-administration
Description: as for outcome 23
Time Frame: Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 276 | 37
minutes | 2.9 (3.96) | 3.8 (2.84)

25. Secondary Outcome: Number of Participants With the Indicated Responses to the Question Regarding the Difficulty of Infusion Site Change
Description: as for outcome 23
Time Frame: Month 12
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 276 | 97
Participants
  Very easy | 143 | 49
  Easy | 130 | 46
  Difficult | 3 | 1
  Very difficult | 0 | 1

26. Secondary Outcome: Number of Participants With the Indicated Responses to the Device Handling Questions
Description: Participants were asked device handling questions to provide information about the impact of the Hylenex administration procedure on everyday life and to investigate perceptions of the overall efficacy and responsiveness of their insulin program. Question 1: Achieve excellent post meal glucose control; Question 2: Insulin responds quickly when basal rate is changed; Question 3: Insulin responds quickly when correction bolus is given.
Time Frame: Month 12
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 276 | 97
Participants
  Question 1: Completely agree | 5 | 0
  Question 1: Agree | 110 | 28
  Question 1: Neither agree or disagree | 97 | 44
  Question 1: Disagree | 59 | 22
  Question 1: Completely disagree | 5 | 3
  Question 2: Completely agree | 31 | 8
  Question 2: Agree | 146 | 48
  Question 2: Neither agree or disagree | 71 | 28
  Question 2: Disagree | 25 | 12
  Question 2: Completely disagree | 3 | 1
  Question 3: Completely agree | 36 | 14
  Question 3: Agree | 165 | 39
  Question 3: Neither agree or disagree | 34 | 22
  Question 3: Disagree | 38 | 20
  Question 3: Completely disagree | 3 | 2

27. Secondary Outcome: Mean Times Per Week Participants Said They Were Eating to Avoid Going Low Due to Late Insulin Action
Description: as for outcome 23
Time Frame: Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: occurrences per week
Arm/Group | Hylenex Recombinant | Standard Rapid-Acting Insulin CSII
Number analyzed (Participants) | 275 | 97
occurrences per week | 2.1 (2.19) | 2.5 (2.37)

ADVERSE EVENTS:
Arm/Group | Commercial Hylenex Recombinant (Formulation 1) | Precommercial Hylenex Recombinant (Formulation 2) | Standard Rapid-Acting Insulin CSII
Serious Adverse Events (participants affected / at risk) | 11/227 | 10/115 | 13/113
Other Adverse Events (participants affected / at risk) | 174/227 | 84/115 | 76/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Commercial Hylenex Recombinant (Formulation 1) (N=227) | Precommercial Hylenex Recombinant (Formulation 2) (N=115) | Standard Rapid-Acting Insulin CSII (N=113)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 3
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1/122 | 0/53 | 0/64
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Stiff person syndrome (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0/122 | 0/53 | 1/64
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Commercial Hylenex Recombinant (Formulation 1) (N=227) | Precommercial Hylenex Recombinant (Formulation 2) (N=115) | Standard Rapid-Acting Insulin CSII (N=113)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 1
Goitre (Endocrine disorders) | 2 | 0 | 0
Hypogonadism (Endocrine disorders) | 1 | 0 | 0
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 1
Conjunctivitis (Eye disorders) | 2 | 0 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 1
Eye discharge (Eye disorders) | 0 | 1 | 0
Macular oedema (Eye disorders) | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 3 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 4 | 0 | 0
Abdominal distention (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 3
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 6 | 2
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 1 | 2
Application site erythema (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 3 | 2 | 1
Feeling hot (General disorders) | 1 | 0 | 0
Infusion site bruising (General disorders) | 5 | 3 | 0
Infusion site discomfort (General disorders) | 0 | 1 | 0
Infusion site erythema (General disorders) | 12 | 4 | 1
Infusion site haematoma (General disorders) | 2 | 0 | 0
Infusion site haemorrhage (General disorders) | 5 | 2 | 0
Infusion site induration (General disorders) | 4 | 0 | 0
Infusion site oedema (General disorders) | 2 | 0 | 0
Infusion site pain (General disorders) | 40 | 17 | 7
Infusion site paraesthesia (General disorders) | 1 | 0 | 0
Infusion site pruritus (General disorders) | 4 | 2 | 0
Infusion site scar (General disorders) | 2 | 0 | 0
Infusion site rash (General disorders) | 1 | 0 | 0
Infusion site reaction (General disorders) | 1 | 1 | 1
Infusion site warmth (General disorders) | 2 | 0 | 0
Injection site pain (General disorders) | 1 | 1 | 0
Injury associated with device (General disorders) | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Oedema peripheral (General disorders) | 3 | 2 | 1
Pyrexia (General disorders) | 1 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 3 | 0 | 0 — The Verbatim term for 1 participant was "Dilantin allergy" and the Verbatim term for the other participant was "Allergic reaction to Keflex and Bactrim".
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 2 | 1 | 0
Abscess oral (Infections and infestations) | 0 | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 2
Atypical pneumonia (Infections and infestations) | 1 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 5 | 5 | 3
Cellulitis (Infections and infestations) | 2 | 0 | 1
Cystitis (Infections and infestations) | 3 | 1 | 1
Ear infection (Infections and infestations) | 5 | 1 | 4
Eye infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 4 | 4 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 5 | 0
Influenza (Infections and infestations) | 6 | 4 | 2
Infusion site infection (Infections and infestations) | 2 | 1 | 1
Kidney infection (Infections and infestations) | 1 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 2 | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Nail infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 26 | 9 | 4
Oral herpes (Infections and infestations) | 1 | 1 | 0
Oral infection (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 1 | 1
Paronychia (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 2
Pharyngitis streptococcal (Infections and infestations) | 1 | 1 | 2
Pneumonia (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 12 | 7 | 8
Skin infection (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 31 | 15 | 13
Urinary tract infection (Infections and infestations) | 10 | 3 | 3
Varicella (Infections and infestations) | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 2 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1 | 2
Concussion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 4 | 0 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Incision cite erythema (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 3 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 2 | 3
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 4 | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0
Fibrin D dimer increased (Investigations) | 1 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 1
Liver function test abnormal (Investigations) | 2 | 0 | 0
Urine ketone body present (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 4 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 2 | 0 | 0
Decreased vibratory sense (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 6 | 2 | 4
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 2
Loss of consciousness (Nervous system disorders) | 0 | 0 | 2
Migraine (Nervous system disorders) | 1 | 1 | 1
Nerve compression (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0
Reflexes abnormal (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Tension headache (Nervous system disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 2 | 2
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 10 | 2 | 1
Insomnia (Psychiatric disorders) | 3 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0 | 0
Pyuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urethral pain (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 0/122 | 1/53 | 0/64
Breast inflammation (Reproductive system and breast disorders) | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1/122 | 0/53 | 1/64
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1/122 | 0/53 | 0/64
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0/122 | 0/53 | 1/64
Uterine polyp (Reproductive system and breast disorders) | 0/122 | 1/53 | 1/64
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 6 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Menopause (Social circumstances) | 1/122 | 0/53 | 0/64
Aortic arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 4 | 1 | 2
Hypotension (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1
Eye haemorrhage (Eye disorders) | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 0
Hunger (General disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1
Allergy to chemicals (Immune system disorders) | 0 | 0 | 1
Allergy to metals (Immune system disorders) | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0
Eye infection viral (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 3 | 1 | 0
H1N1 Influenza (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 2
Hordeolum (Infections and infestations) | 1 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 1
Mycobacteriuim abscessus infection (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fascial rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Carotid bruit (Investigations) | 1 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Tetany (Metabolism and nutrition disorders) | 1 | 0 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Knuckle pads (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 1
Binge eating (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 2 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Wisdom teeth removal (Surgical and medical procedures) | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 0 | 1
Keratitis (Eye disorders) | 1 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information obtained as a result of this study or during the conduct of this study will be regarded as confidential. The Investigator agrees to use the information for the purpose of carrying out this study and for no other purpose, unless written permission from the sponsor (Halozyme) is obtained.